CLINICAL TRIAL: NCT04162730
Title: Validity, Reliability and Responsiveness of Pain Sensitization Questionnaire
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Özgül Öztürk, Principal Investigator, Acibadem University
Other Study IDs: ATADEK 2019/17
Record Dates: First submitted 2019-11-12; First posted 2019-11-14 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Pain Syndrome; Pain, Chronic; Knee Osteoarthritis
MeSH Terms: conditions — Somatoform Disorders; Chronic Pain; Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pressure pain threshold and behavioural data — Pressure pain threshold level of the knee region will be collected and behavioural data will be measured

SUMMARY:
The aim of this study was to translate the Pain Sensitivity Questionnaire, which was developed to determine the level of pain sensitivity of individuals, to Turkish and to evaluate the validity and reliability of the Turkish version of the scale on knee osteoarthritis patients, and as well as to perform cultural adaptation. Pain sensitivity assessment is used to predict treatment or surgical outcomes of individuals. IPain Sensitivity Questionnaire is a frequently used scale that correlates with experimental pain tests and is used in studies conducted in different patient groups. We believe that adding this scale to our language will contribute to other studies in this field.

ELIGIBILITY:
Inclusion Criteria:

* Not having oral or written communication problems in Turkish,
* Diagnosis of knee osteoarthritis after clinical examination and radiological imaging,
* Being 40 years or older,
* To have neurological competence and cognitive level to answer scale questions.

Exclusion Criteria:

* To have fibromyalgia syndrome or neurological disease that may affect pain sensitivity levels of individuals,
* To have undergone surgery involving the knee in the last 1 year,
* The presence of peripheral neuropathy and neuropathy is therefore to be taking medication.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Knee osteoarthritis patients who have chronic pain
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-01-08 (Actual); Primary Completion 2022-12-28 (Estimated); Study Completion 2022-12-28 (Estimated)

PRIMARY OUTCOMES:
Pain Sensitivity Questionnaire | 1-4 week
  The Pain Sensitivity Questionnaire was developed to visualize 17 situations that may feel pain in daily life and to indicate possible pain severity. The patient determines the pain severity level from 0 to 10, with 0 indicates no pain, and 10 indicates the most severe pain. The total score of the Pain Sensitivity Questionnaire and the two subscale scores, PSQ-minor and PSQ-moderate, can be calculated. The PSQ-moderate and PSQ-minor subscales consist of 7 items and the total score is calculated on 14 items. The other 3 items were excluded from the scoring of the scale as they normally indicate painless conditions. Total and subscale scores ranged from 0 to 10, and higher scores indicate increased pain sensitivity.

SECONDARY OUTCOMES:
Pain Catastrophization Scale | 1-4 week
  It consists of a total of 13 items and is scored between 0-52 points. Higher scores mean higher levels of pain catastrophization.
Pressure Pain Threshold | One day

CONTACTS AND LOCATIONS:
Locations (1):
- Özgül Öztürk, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided